CLINICAL TRIAL: NCT04822948
Title: Study of the Intestinal Microbiota During a Real Life Dietary Intervention in Subjects With Overweight or Obesity
Acronym: GUTINSIDE
Status: Completed | Type: Observational
Sponsor: Integrative Phenomics (Industry)
Collaborators: RNPC (Rééducation Nutritionnelle et Psycho-Comportementale) Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: GUT201801
Record Dates: First submitted 2021-03-03; First posted 2021-03-30 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Worldwide, 13% of the population had obesity in 2016 and overweight and obesity are recognized as the fifth leading risk factor for death (roughly 5 million deaths per year). In the United States alone, a recent study predicts that over half of the population will have obesity in 2030. At the global level, overweight and obesity are also estimated to account for 44% of diabetes, 23% of heart disease and between 7% to 41% of cancer cases, in addition to numerous other pathologies, including neurological disorders. While obesity and overweight are classified as a general disease (i.e. a body mass index (BMI) above 25 kg/m2 or 30 kg/m2, respectively), there are large variabilities between classifications of obesity observed. For example, sub-populations of obesity present either a rapid or delayed onset of other chronic diseases, such as diabetes or cardiovascular disease.

Many studies show that lifestyle interventions are effective in improving overweight and obesity through weight loss, but with very large inter-individual variability, especially in the long-term. These interventions and the respective observed weight loss are also shown to reduce the risk of other cardiovascular or metabolic diseases, demonstrating the importance of weight loss for future quality of life Interestingly, there is a large variation in weight loss when implementing the same dietary or lifestyle changes, even when many factors are accounted for in clinical studies. Similar variable weight loss or metabolic responses are also observed for other obesity treatments, such as pharmaceutical or surgical interventions. Therefore, in order to prevent and treat overweight and obesity, it is critical to progress in the understanding of individual variations in responses (trajectories) to weight loss programs.

While biological, environmental, and behavioral factors indeed drive personal responses, recent advances have allowed more insight into how the human body processes these stimuli, namely through microorganisms inhabiting the gastrointestinal tract. Over the last 10 years, the gut microbiota, the 100 billion bacterial cells inhabiting our intestines, has emerged as a recognized factor contributing to our health. Given its access to the food and medicine consumed by an individual, the gut microbiota can be seen as a "super integrator" highly sensitive to our environmental and lifestyle changes. Accumulating evidence has highlighted that the gut microbiota translates these environmental changes by altering its diversity of bacteria or functions and producing molecules that interact with organs and the brain.

As part of a weight loss program conducted within the standard of care in a network of clinical centers across France, the investigators set out to establish a cohort to examine the relative contribution of clinical, nutritional, and lifestyle factors related to individual's weight loss success with an emphasis on evaluating the gut microbiome of individuals.

Within this context, the investigators are testing whether an individuals' microbiota profile before the real-life dietary intervention influences weight loss responses and changes in metabolic health parameters to a standardized weight loss diet.

ELIGIBILITY:
Inclusion Criteria:

* Subject having signed the informed consent
* Male or female, 18 to 65 years of age
* Body Mass Index (BMI) greater than or equal to 25 kg/m²

Exclusion Criteria:

* Pregnant woman (positive serum pregnancy test for selection) or breastfeeding,
* Infected subject under anti-retroviral treatment
* Subject with severe hepatic and / or renal insufficiency (awaiting transplant)
* Subject with anemia <10 g / dl
* Subject with known gastrointestinal illness
* Subject having undergone bariatric surgery
* Subject with a weight loss > 10% of body weight during the last 3 months (special diet: low calorie diet (slimming diet), special diet (vegetarians, vegans, nutritional supplements) before treatment),
* Subject taking pro or prebiotics before treatment
* Subject having taken antibiotics in the 2 months preceding inclusion
* Subject participating in another clinical study,
* Subject not enrolled in the French national healthcare system
* Subject not compliing with the exclusion period from the study in which he/she has previously participated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals who meet the various inclusion criteria as part of the routine care activity of French RNPC centers
Sampling Method: Non-Probability Sample
Enrollment: 1855 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Bodyweight change | 8 weeks
  Bodyweight change calculated relative to baseline body weight

SECONDARY OUTCOMES:
Gut microbiota richness and diversity | Baseline and Estimated: 105 days
  Assessment as gene counts and species
Dietary assessment | Baseline
  Assessment via standardized Food Frequency Questionnaire
Physical activity | Baseline and Estimated: 105 days and 8 months
  Assessment via standardized questionnaire
General health and well-being | Baseline and Estimated: 105 days and 8 months
  Assessment via standardized questionnaire
Eating behavior | Baseline and Estimated: 105 days and 8 months
  Assessment via standardized questionnaire
Body Mass Index (BMI) | Baseline and Estimated: 105 days and 8 months
  Height and bodyweight will be measured to report BMI in (kg/m^2)
Bodyweight | Baseline, Estimated: 105 days and 8 months
  Body weight (kg) measured bi-weekly
Waist circumference | Baseline, Estimated: 105 days and 8 months
  Waist circumference (cm) measured bi-weekly
Body fat mass | Baseline and Estimated: 105 days
  Body fat mass assessed by bioelectrical impedance
Muscle mass | Baseline and Estimated: 105 days
  Muscle mass assessed by bioelectrical impedance
Water weight | Baseline and Estimated: 105 days
  Water weight assessed by bioelectrical impedance
Blood glucose | Baseline and Estimated: 105 days
  Fasting blood glucose
Insulin | Baseline and Estimated: 105 days
  Fasting insulin
HbA1c | Baseline and Estimated: 105 days
  Fasting HbA1c
Blood lipids | Baseline and Estimated: 105 days
  Fasting triglycerides, LDL, HDL
Blood pressure | Baseline and Estimated: 105 days
  Systolic and diastolic blood pressure in mmHg
Liver enzymes | Baseline and Estimated: 105 days
  Fasting levels of AST, ALT, GGT

OTHER OUTCOMES:
Gut microbiota composition | Baseline and Estimated: 105 days
  Assessment of gut microbiota taxonomic features (e.g. phyla, genus, species)

CONTACTS AND LOCATIONS:
Overall Officials: Odile Fabre, Principal Investigator — RNPC
Locations (1):
- RNPC, Marseille, France

IPD SHARING:
Plan to Share IPD: No